CLINICAL TRIAL: NCT02947217
Title: A Randomized Controlled Trial of the Effect of Influenza Vaccination on Implantation and Pregnancy Rates After In-Vitro Fertilization
Brief Title: Effect of Influenza Vaccination on IVF Outcomes - IVF
Acronym: IVF-FluVac
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Center for Human Reproduction (Other)
Collaborators: Foundation for Human Reproduction (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06272016-01 - IVF
Record Dates: First submitted 2016-10-25; First posted 2016-10-27 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Infertility
Keywords: Immunology; Pregnancy; Implantation Rate; Fertilization in Vitro
MeSH Terms: conditions — Infertility | interventions — Influenza Vaccines; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Influenza Vaccine (Experimental): O.5 mL single dose influenza vaccine suspension administered intramuscularly
  Interventions: Biological: Influenza Vaccine
- Saline Injection (Placebo Comparator): O.5 ml of sterile Saline administered intramuscularly
  Interventions: Other: Sterile Saline

INTERVENTIONS:
Biological: Influenza Vaccine — Inactivated influenza vaccine indicated for immunization against disease caused by influenza virus subtype A and type B present in the vaccine. Approved for use in persons 5 years of age and older. Single Dose prefilled 0.5 ml syringe.
  Other Names: Seqirus afluria 2016-2017 formula
  Arms: Influenza Vaccine
Other: Sterile Saline — 0.5 mL of sterile Saline administered im
  Other Names: Saline
  Arms: Saline Injection

SUMMARY:
In this study the investigators propose a randomized controlled trial to evaluate the effect of influenza vaccination on clinical pregnancy rates among women undergoing in vitro fertilization.

DETAILED DESCRIPTION:
Since 2004 flu vaccination has been recommended by American College of Obstetricians and Gynecologists (ACOG) Advisory Committee on Immunization Practices (ACIP) for all pregnant women during flu season, regardless of the trimester of pregnancy. Many studies have examined the safety of influenza vaccination and found benefits beyond the simple prevention of maternal infection including the reduction of still birth. Recently evidence has emerged that women who have received a flu vaccination were less likely to experience premature labor. The investigators hypothesize that some of the maternal benefits of influenza vaccination might be based on other than prevention of the flu, possibly secondary to the induction of immune system pathways that favor immunological tolerance. Induction of immune system pathways that favor immunological tolerance has long been considered a possible path to improved embryo implantation and reduce miscarriages, though the topic is still somewhat controversial.

Patients undergoing IVF will be randomized in two strata:

1. History of recurrent miscarriage or implantation failure
2. No history of recurrent miscarriage of implantation failure

Consenting patients will be randomized to receive either influenza vaccine or a saline placebo. Vaccination will occur 10 days before initiating anticipated menses or fertility treatment cycle start.

All patients will be receiving an offered a second injection at the time of negative pregnancy test or at the time of sign-out with a clinical pregnancy. The second injection will either be placebo or influenza vaccination depending on the original randomization. Patients and clinical staff will remain blinded to the original treatment assignment, except for the study coordinator and the single staff member assigned to administer the injection.

ELIGIBILITY:
Inclusion Criteria:

1. All women preparing to undergo an IVF cycle
2. Women will only be allowed to participate in one treatment cycle
3. Willingness to have an influenza vaccination
4. Signed informed consent

Exclusion Criteria:

1. Any contraindication for flu vaccination
2. Unwillingness to have a flu vaccination
3. Unwillingness to sign informed consent
4. Previous diagnosis of unfavorable endometrial development
5. Unresolved uterine condition that significantly compromises the endometrial cavity

Ages: 21 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Estimated)
Dates: Start 2017-01-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy | 8 weeks
  Intrauterine pregnancy with positive evidence of fetal heart beat

SECONDARY OUTCOMES:
Implantation Rate | 8 weeks
  Number of clinical pregnancies per number of embryos transferred
Evidence of immune activation | 14 to 21 days (at time of egg retrieval)
  Evidence of peripheral markers of immune pathways activated by the influenza vaccine

CONTACTS AND LOCATIONS:
Overall Officials: David H Barad, MD, MS, Principal Investigator — Director of Assisted Reproductive Technology; Norbert Gleicher, MD, Study Director — Medical Director
Locations (1):
- Center For Human Reproduction, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data (IPD)